CLINICAL TRIAL: NCT06525441
Title: The Impact of Dietary Protein Sources on Glycemic Variability in Overweight or Obese Individuals: a Randomized Controlled Trial
Brief Title: Dietary Protein Sources and Glycemic Variability
Acronym: ProG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jie Li, Professor, Deputy director of global health research center, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2024-501-03
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Disease; Diabetes; Overweight; Obesity; Dietary Protein
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus; Overweight; Obesity | interventions — Diet, Plant-Based

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This trial is an open-label study. Given that dietary intervention will be administered to all participants, it is challenging to implement blinding for the participants. However, throughout the study, the individuals involved in the preparation and distribution of meals, along with those conducting the statistical analysis, will remain blind to the group assignments of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plant-based diet (Experimental): Participants assigned to the plant-based diet group will be provided three meals daily for 3 weeks. Of the energy of each meal, 60% is from carbohydrates, 15% from plant protein, and 25% from fat. The main dietary sources of plant protein will be soybeans, flat beans, nuts, grains, and algae.
  Interventions: Other: Plant-based Diet
- Animal-based diet (Active Comparator): Participants assigned to the animal-based diet group will be provided three meals daily for 3 weeks. Of the energy of each meal, 60% is from carbohydrates, 15% from animal protein, and 25% from fat. The main dietary sources of animal protein will be chicken, beef, pork, fish, eggs, and dairy products.
  Interventions: Other: Animal-based Diet

INTERVENTIONS:
Other: Plant-based Diet — Participants assigned to the plant-based diet group will be provided three meals daily for 3 weeks. Of the energy of each meal, 60% is from carbohydrates, 15% from plant protein, and 25% from fat. The main dietary sources of plant protein will be soybeans, flat beans, nuts, grains, and algae.
  Arms: Plant-based diet
Other: Animal-based Diet — Participants assigned to the animal-based diet group will be provided three meals daily for 3 weeks. Of the energy of each meal, 60% is from carbohydrates, 15% from animal protein, and 25% from fat. The main dietary sources of animal protein will be chicken, beef, pork, fish, eggs, and dairy products.
  Arms: Animal-based diet

SUMMARY:
This goal of trial is to evaluate the effects of plant-based vs. animal-based diets on glycemic variability in overweight or obese adults through a 3-week dietary intervention.

The main question it aims to answer is:

Will a plant-based diet be able to reduce glycemic variability in overweight or obese adults compared with an animal-based diet?

Participants will strictly follow a designated plant-based or animal-based dietary regimen throughout the duration of the 3-week study. They will wear a Continuous Glucose Monitor (CGM) throughout the study, engage in weekly clinical assessments, and record their daily dietary intake.

DETAILED DESCRIPTION:
Diabetes stands as one of the most rapidly escalating health challenges of the 21st century. Type 2 diabetes, which represents over 90% of all diagnosed cases, is the predominant form of the disease, with obesity and being overweight identified as key risk factors. The mainstay of prevention and management for Type 2 diabetes continues to be dietary intervention and nutritional therapy. Current dietary strategies for Type 2 diabetes focus predominantly on the regulation of fat and carbohydrate intake, while the influence and underlying mechanisms of dietary protein on glucose metabolism are not yet fully comprehended.

A randomized, open-label, parallel-controlled clinical trial, by strictly controlling the source of protein, will be performed to evaluate the effects of a plant-based diet on glycemic variability and other metabolic outcomes in individuals who are overweight or obese, in comparison to an animal-based diet. Eligible participants will be randomly allocated in a 1:1 ratio to either the plant-based or animal-based diet group for a 3-week intervention.

During the intervention, participants in the plant-based diet group will receive three daily meals for three weeks.Of the energy of each meal, 60% is from carbohydrates, 15% from plant protein, and 25% from fat. The primary sources of plant protein will include soybeans, lentils, nuts, grains, and seaweed. Conversely, the animal-based diet group will also be provided with three daily meals for three weeks, with the same caloric distribution, but sourcing their protein from animal products such as poultry, beef, pork, fish, eggs, and dairy.

Participants are required to cooperate in completing the following tasks:

1. Daily dietary record: Participants are to meticulously track their daily food consumption.
2. Continuous 24-hour glucose monitoring and data logging: Subjects are to undergo continuous monitoring of blood glucose levels throughout a 24-hour period, with all data accurately recorded.
3. Physical examination: This will include assessments of height, weight, waist-to-hip circumference ratio, blood pressure, and body composition.
4. Biological sample collection: Samples to be collected include blood, urine, and stool.

The timing for physical examinations and biological sample collections is scheduled as follows: Day 5 ± 2 of the introduction phase, Week 1 ± 2 days of the intervention phase, Week 2 ± 2 days of the intervention phase, and Week 3 ± 2 days of the intervention phase.

Dietary and health counseling will be consistently available throughout the study to provide participants with continuous support and guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 20-65 years.
2. Body Mass Index (BMI) greater than 25kg/m2.
3. Capable of using a smartphone application daily for taking photos and recording dietary intake.
4. Maintained stable body weight over the past three months with a regular routine.
5. Possess self-care ability for independent living.
6. Not currently participating in any other clinical research projects.
7. Signed the informed consent form and willing to adhere to and complete the entire research process.

Exclusion Criteria:

1. With diagnosed diabetes.
2. With severe cardiovascular or cerebrovascular diseases (e.g., angina, myocardial infarction, or stroke) or cancer.
3. Taking medications affecting weight or energy intake/energy expenditure in the last 3 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician.
4. Participating in weight loss treatments.
5. History of severe gastrointestinal diseases or gastrointestinal surgery within the past 12 months.
6. Those with allergic reactions to common foods (for example, eggs, nuts, grains) or those who are lactose intolerant.
7. Women who are pregnant or plan to become pregnant.
8. Diagnosis of HIV, hepatitis B or C, or active tuberculosis.
9. Special groups who are specifically unsuitable for a diet consisting of whole plant proteins.
10. Patients who are unwilling or unable to give informed consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Amplitude of Glycemic Excursion (MAGE) | From enrollment to the end of intervention at 3 weeks
  Continuous Glucose Monitoring (CGM) will measure the Mean Amplitude of Glycemic Excursion (MAGE).

SECONDARY OUTCOMES:
Change in fasting blood-glucose | From enrollment to the end of intervention at 3 weeks
Change in fasting insulin | From enrollment to the end of intervention at 3 weeks
Change in mean glucose levels | From enrollment to the end of intervention at 3 weeks
Change in total daily time above range | From enrollment to the end of intervention at 3 weeks
  >7.8 mmol/L
Change in total daily time below range | From enrollment to the end of intervention at 3 weeks
  <3.9 mmol/L
Change in range of total daily time | From enrollment to the end of intervention at 3 weeks
  3.9 ~7.8 mmol/L
Change in glycemic variability | From enrollment to the end of intervention at 3 weeks
Change in glycemic standard deviation | From enrollment to the end of intervention at 3 weeks
Change in insulin sensitivity | From enrollment to the end of intervention at 3 weeks
Change in β cell function | From enrollment to the end of intervention at 3 weeks
Change in Large Amplitude of Glycemic Excursions (LAGE) | From enrollment to the end of intervention at 3 weeks
Change in Area Under Curve (AUC) | From enrollment to the end of intervention at 3 weeks
Change in body weight | From enrollment to the end of intervention at 3 weeks
Change in waist-to-hip ratio | From enrollment to the end of intervention at 3 weeks
Change in body composition | From enrollment to the end of intervention at 3 weeks
Change in blood lipids | From enrollment to the end of intervention at 3 weeks
Change in uric acid | From enrollment to the end of intervention at 3 weeks
Change in gut microbiome | From enrollment to the end of intervention at 3 weeks
Change in renal function | From enrollment to the end of intervention at 3 weeks
Change in systolic blood pressure | From enrollment to the end of intervention at 3 weeks
Change in diastolic blood pressure | From enrollment to the end of intervention at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, Principal Investigator — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No